CLINICAL TRIAL: NCT02203032
Title: A Phase 3, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Guselkumab for the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis and an Inadequate Response to Ustekinumab
Brief Title: A Study of Guselkumab in Participants With Moderate to Severe Plaque-type Psoriasis and an Inadequate Response to Ustekinumab
Acronym: NAVIGATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR104918; CNTO1959PSO3003 (Other: Janssen Research & Development, LLC); 2014-000721-20 (EudraCT Number)
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque-type psoriasis; Guselkumab; Ustekinumab; CNTO 1959; Monoclonal antibody
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab; guselkumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-label ustekinumab (Experimental)
  Interventions: Drug: Ustekinumab
- Double-blind guselkumab (Experimental)
  Interventions: Drug: Guselkumab; Drug: Placebo for ustekinumab
- Double-blind ustekinumab (Experimental)
  Interventions: Drug: Ustekinumab; Drug: Placebo for guselkumab

INTERVENTIONS:
Drug: Ustekinumab — 45 mg or 90 mg given by subcutaneous injection at Weeks 0 and 4 for all participants. Participants with an IGA score of 0 or 1 at Week 16 will also receive ustekinumab every 12 weeks (q12w) from Week 16 to Week 40.
  Arms: Double-blind ustekinumab; Open-label ustekinumab
Drug: Guselkumab — 100 mg given by subcutaneous injection at Weeks 16 and 20 and every 8 weeks (q8w) thereafter through Week 44.
  Arms: Double-blind guselkumab
Drug: Placebo for ustekinumab — Subcutaneous injection at Weeks 16, 28, and 40 to maintain the blind for participants randomized to treatment with guselkumab.
  Arms: Double-blind guselkumab
Drug: Placebo for guselkumab — Subcutaneous injection at Weeks 16 and 20 and q8w thereafter through Week 44 to maintain the blind for participants randomized to treatment with ustekinumab.
  Arms: Double-blind ustekinumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of guselkumab (CNTO 1959) in the treatment of participants with moderate to severe plaque-type psoriasis (scaly skin rash) who had inadequate response to ustekinumab.

DETAILED DESCRIPTION:
This is a randomized (assignment of study drug by chance), double-blind (participants nor study staff will know the identity of study drugs), multicenter study to evaluate efficacy and safety of guselkumab for the treatment of participants with moderate to severe plaque-type psoriasis who had an inadequate response to ustekinumab. The study will consist of a screening period, open-label and double-blind treatment periods, and a follow-up period. The treatment period will have 2 phases: an open-label treatment phase during which all participants will receive ustekinumab at Weeks 0 and 4 and a blinded treatment phase during which participants with an inadequate Investigator's Global Assessment response (IGA≥2) to ustekinumab at Week 16 will be randomized to receive either guselkumab or ustekinumab through Week 44. Participants with an IGA response of 0 or 1 (cleared or minimal disease) at Week 16 will continue to receive open-label treatment with ustekinumab every 12 weeks through Week 40. All participants will complete a follow-up phase through Week 52 for efficacy and through Week 60 for safety evaluations. The total duration of the study will be approximately 64 weeks (includes a 4-week screening period). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis (with or without psoriatic arthritis for at least 6 months before the first administration of study drug
* Have a Psoriasis Area and Severity Index (PASI) greater than or equal to (>=) 12 at Screening and at Baseline
* Have an Investigator's Global Assessment (IGA) >=3 at Screening and at Baseline
* Have an involved body surface area (BSA) >= 10 percent (%) at Screening and at Baseline
* Be a candidate for phototherapy or systemic treatment for psoriasis (either naïve or history of previous treatment)

Exclusion Criteria:

* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has unstable cardiovascular disease, defined as a recent clinical deterioration (example [eg], unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months
* Currently has a malignancy or has a history of malignancy within 5 years before Screening (with the exception of a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study drug administration, or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before the first study drug administration)
* Has previously received guselkumab or ustekinumab

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2015-12-25 (Actual); Study Completion 2016-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (85):
- United States (29):
  - Birmingham, Alabama
  - Bakersfield, California
  - Los Angeles, California
  - Santa Monica, California
  - Coral Gables, Florida
  - Ocala, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Skokie, Illinois
  - Indianapolis, Indiana
  - Plainfield, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Troy, Michigan
  - Buffalo, New York
  - New York, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Johnston, Rhode Island
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Webster, Texas
  - Norfolk, Virginia
  - Spokane, Washington
- Australia (4):
  - Fremantle
  - Victoria Park
  - Woden
  - Woolloongabba
- Canada (8):
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - Halifax, Nova Scotia
  - Ajax, Ontario
  - Richmond Hill, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Germany (10):
  - Berlin
  - Bonn
  - Essen
  - Gera
  - Hamburg
  - Leipzig
  - Lübeck
  - Mahlow
  - Münster
  - Witten
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- Russia (7):
  - Chelyabinsk
  - Krasnodar
  - Lipetsk
  - Saint Petersburg
  - Stavropol
  - Ufa
  - Yekaterinburg
- South Korea (3):
  - Anyang
  - Incheon
  - Seoul
- Spain (5):
  - A Coruña
  - Alcorcón
  - Alicante
  - Barcelona
  - Madrid
- Taiwan (4):
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- United Kingdom (4):
  - Dudley
  - Dundee
  - London
  - Salford

REFERENCES:
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Campbell K, Li K, Yang F, Branigan P, Elloso MM, Benson J, Orlovsky Y, Chen Y, Garcet S, Krueger JG. Guselkumab More Effectively Neutralizes Psoriasis-Associated Histologic, Transcriptomic, and Clinical Measures than Ustekinumab. Immunohorizons. 2023 Apr 1;7(4):273-285. doi: 10.4049/immunohorizons.2300003. PMID 37071038

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consists of 2 periods: Open label run-in (Period 1) and blinded phase (Period 2). Participants were enrolled in open label run-in period only. Participants completed the open label run-in period entered into blinded phase period.
Groups:
- Ustekinumab (Open Label Run-in): All participants received ustekinumab 45 milligram (mg) (participants weighing less than or equal to [<=]100 kilogram [kg]) or 90 mg (participants weighing >100 kg) at Weeks 0 and 4. At Week 16, participants with IGA >=2 were randomized to either switch to guselkumab 100 mg at Weeks 16 and 20 and then every 8 weeks thereafter or continue on ustekinumab every 12 weeks (q12w); participants with an IGA=0 or 1 were to continue to receive open-label ustekinumab q12w.
- 100 mg Guselkumab (Randomized): Participants from open label run-in phase with an investigator global assessment (IGA) greater than or equal to (>=) 2 at Week 16 who were randomized to guselkumab, received guselkumab 100 mg at Weeks 16, 20, 28, 36, and 44 and placebo for ustekinumab at Weeks 16, 28, and 40.
- Ustekinumab (Randomized): Participants from open label run-in phase with an IGA >=2 at Week 16 who were randomized to ustekinumab, continued to receive ustekinumab, according to their baseline (Week 0) weight, at Weeks 16, 28, and 40, and placebo for guselkumab at Weeks 16, 20, 28, 36, and 44.
- Ustekinumab (Nonrandomized Open Label Continuation): Participants from open label run-in phase with an IGA=0 or 1 at Week 16 received ustekinumab 45 mg or 90 mg (according to their baseline weight [Week 0]) at Weeks 16, 28, and 40.
Period: Open Label Run-in (Week 0 to Week 16)
Arm/Group | Ustekinumab (Open Label Run-in) | 100 mg Guselkumab (Randomized) | Ustekinumab (Randomized) | Ustekinumab (Nonrandomized Open Label Continuation)
Started | 872 | 0 | 0 | 0
Treated | 871 | 0 | 0 | 0
Completed | 853 | 0 | 0 | 0
Not Completed | 19 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0
Not completed — Enrolled but not treated | 1 | 0 | 0 | 0
Period: Blinded Phase (Week 16 to Week 44)
Arm/Group | Ustekinumab (Open Label Run-in) | 100 mg Guselkumab (Randomized) | Ustekinumab (Randomized) | Ustekinumab (Nonrandomized Open Label Continuation)
Started | 0 | 135 | 133 | 585
Completed | 0 | 120 | 107 | 539
Not Completed | 0 | 15 | 26 | 46
Not completed — Lost to Follow-up | 0 | 2 | 3 | 8
Not completed — Withdrawal by Subject | 0 | 8 | 19 | 20
Not completed — Other | 0 | 4 | 1 | 15
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Completed Safety follow-up | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis included all participants who were enrolled at Week 0 and received at least 1 dose of study agent administration.
Arm/Group | Ustekinumab (Open Label Run-in)
Number analyzed (Participants) | 871
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 814
  >=65 years | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305
  Male | 566
Region of Enrollment [Number; unit: participants]
  Germany | 96
  Poland | 294
  Russia | 88
  Spain | 24
  United Kingdom | 11
  Canada | 61
  United States | 194
  Australia | 19
  Korea, Republic Of | 29
  Taiwan, Province Of China | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Visits at Which Participants Achieved an Investigator's Global Assessment (IGA) Response of Cleared (0) or Minimal (1) and at Least a 2 Grade Improvement (From Week 16) From Week 28 Through Week 40
Description: The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 28 through Week 40
Population: Randomized population included all enrolled participants with IGA >=2 at Week 16 randomly assigned to 1 of the 2 treatment regimens (guselkumab or ustekinumab) at Week 16.
Measure: Mean (Standard Deviation); unit: visits
Groups:
- Guselkumab (Randomized): Participants from open label Run-in phase with an investigator global assessment (IGA) greater than or equal to (>=) 2 at Week 16 who were randomized to guselkumab, received guselkumab 100 mg at Weeks 16, 20, 28, 36, and 44 and placebo for ustekinumab at Weeks 16, 28, and 40.
Arm/Group | Guselkumab (Randomized) | Ustekinumab (Randomized)
Number analyzed (Participants) | 135 | 133
visits | 1.5 (1.57) | 0.7 (1.26)
Statistical Analysis 1: Comparison: Guselkumab (Randomized) vs Ustekinumab (Randomized); Test type: Superiority or Other; p < 0.001, Row mean score test

2. Secondary Outcome: Number of Visits at Which Participants Achieved a Psoriasis Area and Severity Index (PASI) 90 Response From Week 28 Through Week 40
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Time Frame: Week 28 through Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Guselkumab (Randomized) | Ustekinumab (Randomized)
Number analyzed (Participants) | 135 | 133
visits | 2.2 (1.69) | 1.1 (1.53)
Statistical Analysis 1: Comparison: Guselkumab (Randomized) vs Ustekinumab (Randomized); Test type: Superiority or Other; p < 0.001, Row mean score test

3. Secondary Outcome: Number of Visits at Which Participants Achieved an IGA Score of Cleared (0) From Week 28 Through Week 40
Description: as for outcome 1
Time Frame: Week 28 through Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Guselkumab (Randomized) | Ustekinumab (Randomized)
Number analyzed (Participants) | 135 | 133
visits | 0.9 (1.34) | 0.4 (1.06)
Statistical Analysis 1: Comparison: Guselkumab (Randomized) vs Ustekinumab (Randomized); Test type: Superiority or Other; p < 0.001, Row mean score test

4. Secondary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) and at Least a 2 Grade Improvement (From Week 16) at Week 28
Description: as for outcome 1
Time Frame: Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab (Randomized) | Ustekinumab (Randomized)
Number analyzed (Participants) | 135 | 133
percentage of participants | 31.1 | 14.3
Statistical Analysis 1: Comparison: Guselkumab (Randomized) vs Ustekinumab (Randomized); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Up to Week 60
Description: Safety analysis included all participants who were enrolled at Week 0 and received at least 1 dose of study agent administration.
Arm/Group | Ustekinumab (Open Label Run-in) | 100 mg Guselkumab (Randomized) | Ustekinumab (Randomized) | Ustekinumab (Nonrandomized Open Label Continuation)
Serious Adverse Events (participants affected / at risk) | 11/871 | 9/135 | 6/133 | 20/585
Other Adverse Events (participants affected / at risk) | 80/871 | 37/135 | 33/133 | 60/585
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab (Open Label Run-in) (N=871) | 100 mg Guselkumab (Randomized) (N=135) | Ustekinumab (Randomized) (N=133) | Ustekinumab (Nonrandomized Open Label Continuation) (N=585)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Sinus Node Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 2
Retinal Artery Embolism (Eye disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Paraspinal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Scapula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab (Open Label Run-in) (N=871) | 100 mg Guselkumab (Randomized) (N=135) | Ustekinumab (Randomized) (N=133) | Ustekinumab (Nonrandomized Open Label Continuation) (N=585)
Nasopharyngitis (Infections and infestations) | 47 | 23 | 23 | 33
Upper Respiratory Tract Infection (Infections and infestations) | 33 | 15 | 11 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.